CLINICAL TRIAL: NCT03669263
Title: Fentanyl Buccal Soluble Films Feasible Dose Range Study for Breakthrough Pain in Taiwanese Cancer Patients
Brief Title: A Dose Titration Study of Fentanyl Buccal Soluble Film for Breakthrough Cancer Pain in Taiwan
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: TTY Biopharm (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PK1302
Record Dates: First submitted 2018-08-17; First posted 2018-09-13 (Actual); Last update posted 2018-09-13 (Actual); Status verified 2018-08

CONDITIONS: Breakthrough Cancer Pain
Keywords: Painkyl®; fentanyl buccal soluble film; dose titration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Fentanyl buccal soluble film (FBSF) (Experimental): Single arm
  Interventions: Drug: Fentanyl buccal soluble film (FBSF)

INTERVENTIONS:
Drug: Fentanyl buccal soluble film (FBSF) — After screening, eligible subjects were individually titrated to an adequate dose of FBSF (titration period) and continued on this dose as required to control their BTP throughout the maintenance period of the study.
  During the dose titration period, subjects were administered with FBSF in a dose escalation manner until a treatment dose was identified (defined as an adequate relief of BTP observed for at least two consecutive episodes). All patient started with a dose of 200 μg and increased by 200 μg in each subsequent episode until an adequate pain relief with tolerable side effects was achieved. Doses above 1200 μg were not allowed.
  Other Names: Painkyl, fentanyl buccal soluble film (FBSF)

SUMMARY:
Primary Objective:

To determine the feasible dose range of Painkyl® required for Taiwanese population.

Secondary Objectives:

To evaluate the efficacy of Painkyl® by calculating squared mean of pain intensity difference at 30 minutes after taking Painkyl® (SPID30, an 11-point scale).

To evaluate subjects' satisfaction by conducting global evaluation of medication performance (a 5-point categorical scale).

To identify percentage of episodes requiring rescue medication during maintenance treatment period.

To evaluate the safety data of Painkyl® for breakthrough pain.

DETAILED DESCRIPTION:
The primary endpoint was the feasible range of FBSF required for Taiwanese population. The secondary endpoints were the difference in pain intensity at 30 minutes (PID30) after FBSF administration, subjects' satisfaction, and the percentage of episodes requiring rescue medications.

Pain intensity was determined using an 11-point numeric scale from 0="no pain" to 10="worst pain." Patients were assessed with baseline pain as well as pain intensity at 30 minutes after dosing. The PID30 was obtained by baseline pain score minus score rated 30 minutes after dosing.

Patient's satisfaction was assessed using a 5-point (poor, fair, good, very good, and excellent) categorical scale at 30 minutes after taking FBSF with the following question: "What was your overall satisfaction with the medication?" At each episode of BTP, subjects recorded whether a rescue medication was taken after administration of FBSF.

ELIGIBILITY:
Inclusion Criteria:

* a. a stable current regimen of oral opioids equivalent to 60-1000 mg/day of oral morphine or 20-120 mg/day of iv morphine or 25-300 mcg/hr of transdermal fentanyl for one week or longer;
* b. regularly experienced 1 to 3 breakthrough pain episodes per day that required additional opioids from pain control;
* c. at least partial relief of breakthrough pain by use of opioid therapy;
* d. 20 years of age or older;
* e. ability to understand and willingness to sign a written informed consent document;
* f. able to self-administer the study medication correctly or has the availability of a responsible adult caregiver available to administer the study medication correctly;
* g. willing and able to complete patient diary with each pain episode

Exclusion Criteria:

* a. rapidly escalating pain (e.g., regularly more than 3 breakthrough pain episodes per day) that are hard to be controlled by analgesics;
* b. history of hypersensitivity or intolerance to fentanyl;
* c. cardiopulmonary disease that, in the opinion of the investigator, would significantly increase the risk of respiratory depression;
* d. psychiatric/cognitive or neurological impairment that would limit the subject's ability to understand or complete the diary;
* e. moderate (Grade 3) to severe (Grade 4) mucositis (subjects with less than moderate mucositis are permitted and must be instructed to not apply the Painkyl® film at a site of inflammation);
* f. abnormal oral mucosa which will impede drug absorption;
* g. currently under other treatments that may alter effect of pain control based on investigator's judgment;
* h. recent history or current evidence of alcohol or other drug substance (licit or illicit) abuse;
* i. use of an investigational drug within 4 weeks preceding this study;
* j. pregnant women or nursing mothers, or positive pregnancy test for women of childbearing potential;

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-11-25 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2016-07-01 (Actual)

PRIMARY OUTCOMES:
Optimal dose calculation of Painkyl® | Within 2 weeks
  Time to "optimal" dose of an open-label study medication in the titration phase. During the dose titration period, subjects were administered with FBSF (Painkyl®) in a dose escalation manner until a treatment dose was identified (defined as an adequate relief of BTP observed for at least two consecutive episodes). All patient started with a dose of 200 μg and increased by 200 μg in each subsequent episode until an adequate pain relief with tolerable side effects was achieved.

SECONDARY OUTCOMES:
Efficacy Phase : Pain intensity difference at 30 minutes (PID30) after treatment | During the efficacy phase, at each episode of breakthrough pain, 30 minutes after taking dose of study drug, at 0 and 10 minutes after taking dose of study drug
  During the efficacy phase participants assessed their pain intensity at each breakthrough pain (BTP) episode at 0 and 30 minutes after taking dose using the 11-point Numerical Rating Scale (NRS) on a scale from 0 to 10, where 0 represents the absence of pain and 10 is "worst possible pain". PID30 is calculated as the difference in pain intensity from time 0 to 30 minutes. A positive value is a decrease (improvement) of the pain; a ≥ 3-point difference is considered as clinically important.
Efficacy Phase : Subjects' satisfaction score at 30 minutes after treatment | During the efficacy phase, at each episode of breakthrough pain, 30 minutes after taking dose of study drug
  Participants assessed their subjects' satisfaction of treatment efficacy for treated BTP episodes at 30 minutes after taking dose of study drug. The validated, categorical 5-point Verbal Rating Scale (VRS) was used for this assessment and scored as follows: poor; fair; good; very good; excellent.
The percentage of episodes requiring rescue medications. | Within 2 weeks
  • Percentage of episodes requiring rescue medications: subjects will record whether rescue medication was taken after study medication administration for each episode of BTP, by answering "yes" or "no."
Incidence of adverse events (AEs), serious adverse events (SAEs) [Safety and Tolerability] | From the date of study entry until 30 days after the last dose of study treatment
  Assessed by the NCI-CTCAE (Common Toxicity Criteria for Adverse Effects) v4.0 and within some subgroups of patients

CONTACTS AND LOCATIONS:
Overall Officials: Cheng-Hsu Wang, Study Chair — Chang Gung Memorial Hospital, Linkou, Taiwan
Locations (1):
- Chang Gung Memorial Hospital, Keelung, Taiwan

REFERENCES:
- [Background] Greco MT, Corli O, Montanari M, Deandrea S, Zagonel V, Apolone G; Writing Protocol Committee; Cancer Pain Outcome Research Study Group (CPOR SG) Investigators. Epidemiology and pattern of care of breakthrough cancer pain in a longitudinal sample of cancer patients: results from the Cancer Pain Outcome Research Study Group. Clin J Pain. 2011 Jan;27(1):9-18. doi: 10.1097/AJP.0b013e3181edc250. PMID 20842024
- [Background] Rhiner MI, von Gunten CF. Cancer breakthrough pain in the presence of cancer-related chronic pain: fact versus perceptions of health-care providers and patients. J Support Oncol. 2010 Nov-Dec;8(6):232-8. doi: 10.1016/j.suponc.2010.10.006. PMID 21265388
- [Background] Mercadante S. The use of rapid onset opioids for breakthrough cancer pain: the challenge of its dosing. Crit Rev Oncol Hematol. 2011 Dec;80(3):460-5. doi: 10.1016/j.critrevonc.2010.12.002. Epub 2011 Jan 6. PMID 21215653
- [Background] Rauck R, North J, Gever LN, Tagarro I, Finn AL. Fentanyl buccal soluble film (FBSF) for breakthrough pain in patients with cancer: a randomized, double-blind, placebo-controlled study. Ann Oncol. 2010 Jun;21(6):1308-1314. doi: 10.1093/annonc/mdp541. Epub 2009 Nov 25. PMID 19940014
- [Derived] Chiou TJ, Chao TC, Chao TY, Huang JS, Chang YF, Wang CH. A dose titration study of fentanyl buccal soluble film for breakthrough cancer pain in Taiwan. Cancer Rep (Hoboken). 2019 Oct;2(5):e1179. doi: 10.1002/cnr2.1179. Epub 2019 Apr 23. PMID 32721110